CLINICAL TRIAL: NCT03186820
Title: Exploratory Study of the Interest of MRI Susceptibility Weighted Imaging for the Pre-operative Assessment of Pelvic Endometriosis Extent
Acronym: EndoSWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2017/03
Record Dates: First submitted 2017-06-02; First posted 2017-06-14 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; Magnetic resonance imaging (MRI); Susceptibility-weighted imaging (SWI)
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Prospective monocentric comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SWAN sequence (Experimental): Susceptibility Weighted Imaging as 3D SWAN sequence
  Interventions: Other: Susceptibility Weighted Imaging as 3D SWAN sequence

INTERVENTIONS:
Other: Susceptibility Weighted Imaging as 3D SWAN sequence — Susceptibility Weighted Imaging as 3D SWAN sequence

SUMMARY:
Knowledge of the precise location of endometriosis is essential for a successful surgical treatment. MRI Susceptibility-Weighted Imaging (SWI-MRI) yields high sensitivity for blood by-products detection. Since endometriosis lesions are haemorrhagic, and therefore rich in blood by-products such as hemosiderin, SWI-MRI could be useful in the pre-operative assessment of endometriosis, especially in superficial peritoneal lesion detection. The purpose of our study is to evaluate the performance of SWI-MRI for the preoperative work-up of endometriosis

DETAILED DESCRIPTION:
Pelvic endometriosis is a cause of pelvic pain, dysmenorrhea, urinary symptoms and infertility. MRI is considered as the best imaging technique to detect and to predict the extent of the disease. Susceptibility Weighted Imaging is routinely performed to identify haemorrhagic lesions in brain MRI protocols and has proven to be a sensitive technique to detect blood by-products. A pelvic MRI protocol including SWI will be performed in all women addressed for diagnostic assessment or pre-operative work-up of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (over 18yrs old) addressed for diagnostic assessment or pre-operative work-up of endometriosis;
* Informed signed consent
* Affiliated or beneficiary of a social security system

Exclusion Criteria:

* Patient <18yrs old
* Pregnant or nursing woman
* Patient under legal protection
* Contraindication to MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Interest of MRI Susceptibility Weighted Imaging | Baseline (MRI) and day of surgery
  The diagnostic use of SWI-MRI will be assessed through:
  * the number of endometriotic locations, which are both identified with SWI-MRI and confirmed by surgery.
  * the sensitivity, specificity, and predictive values of MRI.
  * signal intensities of each endometriotic location found in surgery on T1 weighted sequence (presence of a high signal intensity) and SWI (presence of a low signal intensity)

SECONDARY OUTCOMES:
Deep forms of endometriosis | Baseline (MRI) and day of surgery
  MRI findings will be compared to surgical findings
Superficial forms of endometriosis | Baseline (MRI) and day of surgery
  MRI findings will be compared to surgical findings

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saha R, Kuja-Halkola R, Tornvall P, Marions L. Reproductive and Lifestyle Factors Associated with Endometriosis in a Large Cross-Sectional Population Sample. J Womens Health (Larchmt). 2017 Feb;26(2):152-158. doi: 10.1089/jwh.2016.5795. Epub 2016 Sep 15. PMID 27632570
- [Background] Olive DL, Schwartz LB. Endometriosis. N Engl J Med. 1993 Jun 17;328(24):1759-69. doi: 10.1056/NEJM199306173282407. No abstract available. PMID 8110213
- [Background] Siegelman et al." Radiographics: A Review Publication of the Radiological Society of North America, Inc 32, no. 6 (October 2012).
- [Background] Fritzer N, Haas D, Oppelt P, Renner S, Hornung D, Wolfler M, Ulrich U, Fischerlehner G, Sillem M, Hudelist G. More than just bad sex: sexual dysfunction and distress in patients with endometriosis. Eur J Obstet Gynecol Reprod Biol. 2013 Jul;169(2):392-6. doi: 10.1016/j.ejogrb.2013.04.001. Epub 2013 May 1. PMID 23642970
- [Background] Chapron C, Dubuisson JB. Management of deep endometriosis. Ann N Y Acad Sci. 2001 Sep;943:276-80. doi: 10.1111/j.1749-6632.2001.tb03808.x. PMID 11594547
- [Background] Benacerraf BR, Groszmann Y. Sonography should be the first imaging examination done to evaluate patients with suspected endometriosis. J Ultrasound Med. 2012 Apr;31(4):651-3. doi: 10.7863/jum.2012.31.4.651. No abstract available. PMID 22441923
- [Background] Holland TK, Cutner A, Saridogan E, Mavrelos D, Pateman K, Jurkovic D. Ultrasound mapping of pelvic endometriosis: does the location and number of lesions affect the diagnostic accuracy? A multicentre diagnostic accuracy study. BMC Womens Health. 2013 Oct 29;13:43. doi: 10.1186/1472-6874-13-43. PMID 24165087
- [Background] Abrao et al. "Comparison between Clinical Examination, Transvaginal Sonography and Magnetic Resonance Imaging for the Diagnosis of Deep Endometriosis." Human Reproduction (Oxford, England) 22, no. 12 (December 2007). Bazot et al. "Diagnostic Accuracy of Physical Examination, Transvaginal Sonography, Rectal Endoscopic Sonography, and Magnetic Resonance Imaging to Diagnose Deep Infiltrating Endometriosis." Fertility and Sterility 92, no. 6 (December 2009). Bazot, M., N. Bharwani, C. Huchon, K. Kinkel, T. M. Cunha, A. Guerra, L. Manganaro, et al. "European Society of Urogenital Radiology (ESUR) Guidelines: MR Imaging of Pelvic Endometriosis." European Radiology, December 5, 2016
- [Background] Jarlot C, Anglade E, Paillocher N, Moreau D, Catala L, Aube C. [MR imaging features of deep pelvic endometriosis: correlation with laparoscopy]. J Radiol. 2008 Nov;89(11 Pt 1):1745-54. doi: 10.1016/s0221-0363(08)74479-2. French. PMID 19106831
- [Background] Bazot M, Gasner A, Lafont C, Ballester M, Darai E. Deep pelvic endometriosis: limited additional diagnostic value of postcontrast in comparison with conventional MR images. Eur J Radiol. 2011 Dec;80(3):e331-9. doi: 10.1016/j.ejrad.2010.12.006. Epub 2011 Jan 7. PMID 21216125
- [Background] Siegelman ES, Oliver ER. MR imaging of endometriosis: ten imaging pearls. Radiographics. 2012 Oct;32(6):1675-91. doi: 10.1148/rg.326125518. PMID 23065164
- [Background] Siegelman ES, Outwater E, Wang T, Mitchell DG. Solid pelvic masses caused by endometriosis: MR imaging features. AJR Am J Roentgenol. 1994 Aug;163(2):357-61. doi: 10.2214/ajr.163.2.8037030.
- [Background] Haacke EM, Mittal S, Wu Z, Neelavalli J, Cheng YC. Susceptibility-weighted imaging: technical aspects and clinical applications, part 1. AJNR Am J Neuroradiol. 2009 Jan;30(1):19-30. doi: 10.3174/ajnr.A1400. Epub 2008 Nov 27. PMID 19039041
- [Background] Nair JR, Van Hecke W, De Belder F, Venstermans C, van den Hauwe L, Van Goethem J, Parizel PM. High-resolution susceptibility-weighted imaging at 3 T with a 32-channel head coil: technique and clinical applications. AJR Am J Roentgenol. 2010 Oct;195(4):1007-14. doi: 10.2214/AJR.10.4218. PMID 20858832
- [Background] Bai Y, Wang MY, Han YH, Dou SW, Lin Q, Guo Y, Li W, Ding DG, Dai JP, Qin W, Shi DP, Tian J, Dai YM. Susceptibility weighted imaging: a new tool in the diagnosis of prostate cancer and detection of prostatic calcification. PLoS One. 2013;8(1):e53237. doi: 10.1371/journal.pone.0053237. Epub 2013 Jan 7. PMID 23308170
- [Background] Cimsit C, Yoldemir T, Guclu M, Akpinar IN. Susceptibility-weighted magnetic resonance imaging for the evaluation of deep infiltrating endometriosis: preliminary results. Acta Radiol. 2016 Jul;57(7):878-85. doi: 10.1177/0284185115602147. Epub 2015 Aug 27. PMID 26315838
- [Background] Takeuchi M, Matsuzaki K, Harada M. Susceptibility-weighted MRI of extra-ovarian endometriosis: preliminary results. Abdom Imaging. 2015 Oct;40(7):2512-6. doi: 10.1007/s00261-015-0378-z. PMID 25682291
- [Background] Takeuchi M, Matsuzaki K, Nishitani H. Susceptibility-weighted MRI of endometrioma: preliminary results. AJR Am J Roentgenol. 2008 Nov;191(5):1366-70. doi: 10.2214/AJR.07.3974. PMID 18941070
- [Background] Solak A, Sahin N, Genc B, Sever AR, Genc M, Sivrikoz ON. Diagnostic value of susceptibility-weighted imaging of abdominal wall endometriomas during the cyclic menstrual changes: a preliminary study. Eur J Radiol. 2013 Sep;82(9):e411-6. doi: 10.1016/j.ejrad.2013.04.030. Epub 2013 Jun 10. PMID 23763857